CLINICAL TRIAL: NCT06845397
Title: Chuvashia Inappropriate Prescribing Study
Acronym: CHIP
Status: Completed | Type: Observational
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Collaborators: BU "Respublikanski Kardiologicheski Dispanser" Minzdrava Chuvashii, Cheboksary (Unknown)
Responsible Party: Sponsor
Other Study IDs: 06-07/23
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Multimorbidity, Cardiovascular Diseases
Keywords: multimorbidity; self-medication; drugs; over-the-counter (OTC) drugs; prescription drugs; adherence; inappropriate prescribing
MeSH Terms: conditions — Cardiovascular Diseases; Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a cross-sectional study based on an outpatient registry. All medical therapy will be registered in order to assess inappropriate prescribing's, in accordance with the criteria PROMPT and BEERS, also in accordance with the officially approved instructions for the use of this medicinal product.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years old, multimorbidity, signed Patients' Informed Consent

Exclusion Criteria:

* Age < 50 years, presence of mental illnesses, oncological diseases detected less than 5 years ago, acute cardiovascular pathology within 6 months prior to inclusion.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a cross-sectional study based on an outpatient registry. All medical therapy will be registered in order to assess inappropriate prescribing's, in accordance with the criteria PROMPT and BEERS, also in accordance with the officially approved instructions for the use of this medicinal product.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
frequency of inappropriate drug prescriptions | Assessed at baseline
  Рrescribing medications in an inadequate dose, with the wrong frequency, and the wrong duration of treatment, failure to prescribe a potentially effective drug in the presence of clinical indications, self-medication was considered irrational treatment and was assessed as the end point.
  It also includes prescribing medications that are likely to have a negative effect on the course of concomitant pathology, as well as drug interactions, in accordance with the criteria PROMPT and BEERS.

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Martsevich, M.D., Professor, Study Director — National Medical Research Centre for Therapy and Preventive Medicine, Moscow, Russia
Locations (1):
- Respublikanski Kardiologicheski Dispanser Minzdrava Chuvashii, Cheboksary, Russia

IPD SHARING:
Plan to Share IPD: No